CLINICAL TRIAL: NCT05208697
Title: Tele-Harm Reduction for Rapid Initiation of Antiretrovirals in People Who Inject Drugs: a Randomized Controlled Trial
Brief Title: Tele-Harm Reduction
Acronym: T-SHARP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Hansel Tookes, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20201516; DP2DA053720 (NIH)
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: IV Drug Usage; HIV Infections; Hepatitis C
Keywords: heroin; needle exchange; syringe services program
MeSH Terms: conditions — HIV Infections; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Harm Reduction (THR) (Experimental): THR utilizes 2 components. Component 1: telehealth technology facilitated by a peer harm reduction counselor to connect the participant with medical case managers and enroll patients in Ryan White/AIDS Drug Assistance Program (ADAP). Component 2: utilizes the syringe services program (SSP)-based peer harm reduction counselor to work with participants in identifying individual-specific barriers and facilitators to medication adherence.
  Interventions: Behavioral: Tele-Harm Reduction
- off-site linkage to HIV care (Active Comparator): introduces the participant to an SSP HIV/HCV linkage specialist and discusses linkage to a traditional Ryan White clinic
  Interventions: Other: off-site linkage

INTERVENTIONS:
Behavioral: Tele-Harm Reduction — THR is telehealth-enhanced, on-demand services including low-barrier access to antiretrovirals, medications for substance use disorder and hepatitis C treatment. It includes mobile phlebotomy, harm reduction counseling, medication management, telehealth mental health/substance use disorder services-- all delivered via an SSP, integrated with the provision of evidence-based naloxone and injection equipment.
  Arms: Tele-Harm Reduction (THR)
Other: off-site linkage — standard of care linkage to a Ryan White clinic
  Arms: off-site linkage to HIV care

SUMMARY:
The purpose of this study is to test 2 different methods for offering medications that treat HIV, cure Hepatitis C Virus (HCV) (if applicable) and treat substance use disorder (if desired) to people who inject drugs.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* able to speak English
* enrolled in IDEA Miami or IDEA Tampa SSPs
* injection drug use in past 12 months by self-report
* willing and able to sign informed consent, provide locator information and medical records release
* testing reactive for HIV by rapid test
* HIV RNA>200 copies/ml as determined by on-site labs or abstracted medical records (result within 3 months of randomization date)

Exclusion Criteria:

* testing HIV negative via rapid test
* receipt of THR intervention in the past 6 months
* inability to provide informed consent
* planning to leave the area within 12 months
* Principal or site investigator discretion
* currently in prison or jail
* Enrollment in Clinical Trials Network 121

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Viral suppression | up to 12 months
  HIV viral load <200 copies/ml time-averaged

SECONDARY OUTCOMES:
Initiation of medications for opioid use disorder | up to 12 months
  Positive urine drug screen for buprenorphine, naltrexone or methadone at study follow-up visit after MOUD is prescribed.
HCV cure | up to 12 months
  HCV treatment initiated resulting in negative HCV RNA at 12 weeks post treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Hansel Tookes, MD, MPH, Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - Care Resource The SPOT, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tookes HE, Oxner A, Serota DP, Alonso E, Metsch LR, Feaster DJ, Ucha J, Suarez E Jr, Forrest DW, McCollister K, Rodriguez A, Kolber MA, Chueng TA, Zayas S, McCoy B, Sutherland K, Archer C, Bartholomew TS. Project T-SHARP: study protocol for a multi-site randomized controlled trial of tele-harm reduction for people with HIV who inject drugs. Trials. 2023 Feb 7;24(1):96. doi: 10.1186/s13063-023-07074-w. PMID 36750867